CLINICAL TRIAL: NCT01930331
Title: Safety, Tolerability, Pharmacokinetics and Efficacy, Phase Iv, Open Label Study of Fixed Arco® and Eurartesim® Therapies in Adults and Children With Uncomplicated P. Falciparum Malaria in Tanzania
Brief Title: Safety, Tolerability, Pharmacokinetics and Efficacy of ARCO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ifakara Health Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IHI
Record Dates: First submitted 2013-08-09; First posted 2013-08-28 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Plasmodium Falciparum; Malaria, Falciparum
Keywords: Uncomplicated Plasmodium falciparum Malaria
MeSH Terms: conditions — Malaria, Falciparum | interventions — artemisinin; naphthoquine; artemisinin-naphthoquine combination; artenimol; piperaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ARCO treatment (Experimental): Patients in this treatment arm will receive on Day 0 a single dose of standard treatment of artemisinin/naphthoquine (in a fixed oral dose of ARCO tablets). Treatment will be given under supervision.
  Interventions: Drug: artemisinin/naphthoquine
- Eurartesim treatment (Active Comparator): Patients in this treatment arm will receive a dose of dihydroartemisinin/piperaquine phosphate (in a fixed oral dose of Eurartesim tablets) over three days (0,1,2). Treatment will be given under supervision.
  Interventions: Drug: dihydroartemisinin/piperaquine phosphate

INTERVENTIONS:
Drug: artemisinin/naphthoquine — Each tablet of ARCO (artemisinin/naphthoquine) contains 125 mg artemisinin and 50 mg of naphthoquine. The total dose for adults will be 1000mg of artemisinin and 400mg of naphthoquine in a fixed oral dose (ARCO tablet).
  The regimen for children will be calculated according to the body weight (20mg artemisinin + 8mg naphthoquine per kg body weight in a fixed oral dose(ARCO tablet)).
  Other Names: ARCO®
  Arms: ARCO treatment
Drug: dihydroartemisinin/piperaquine phosphate — Eurartesim (dihydroartemisinin/piperaquine phosphate) is a fixed dose preparation with two dose-strengths (20 mg dihydroartemisinin and 160mg of piperaquine phosphate and 40mg dihydroartemisinin and 320mg of piperaquine phosphate. The regimen for patients with body weight of 36-75kg is three tablets of 40mg dihydroartemisinin and 320mg of piperaquine phosphate once daily for three consecutive days. Those beyond or below this range the regimen will be calculated based on the body weight.
  Other Names: Eurartesim®
  Arms: Eurartesim treatment

SUMMARY:
Phase IV, single center, 2 arms randomized controlled, open label study. Study will be conducted over a period of 42 days to determine the safety, tolerability, pharmacokinetics and efficacy of ARCO.

DETAILED DESCRIPTION:
Evaluation of safety and tolerability of the administration of ARCO and Eurartesim in terms of blood biochemistry, full blood count, ECG assessments, vital signs and adverse events profile in patients with uncomplicated P. falciparum malaria. Dihydroartemisinin/piperaquine will be used as comparator.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent, in accordance with local practice, provided by patient, for children it will provided by either parents or legal representative and in addition children will provide assent.
2. Male or female patients between the age of 6 and 60 years (both inclusive)
3. Body weight between 20 kg and 90 kg (both inclusive)
4. Presence of mono-infection with P. falciparum (1,000 to 100,000 asexual count/µl of blood) microscopically confirmed.
5. Fever, as defined by axillary temperature ≥ 37.5°C to ≤ 39.5°C
6. Ability to swallow oral medication
7. Ability and willingness to adhere to all study procedures and access health facilities.
8. Agree to undergo study related procedures including being hospitalized for minimum of 3 days (0,1 and 2), and a follow up of up to 42 days.

Exclusion Criteria:

1. Patients with signs and symptoms of severe/complicated malaria as described in the WHO guideline(Third Edition 2012) for management of severe malaria(6)(Appendix 1)
2. Mixed Plasmodial infection.
3. Severe vomiting, defined as more than three times in the 24 hours prior to inclusion in the study or inability to tolerate oral treatment.
4. Severe diarrhoea defined as 3 or more watery stools per day.
5. Presence of other serious or chronic clinical condition requiring hospitalization.
6. Known history or evidence of clinically significant disorders such as cardiovascular (including arrhythmia, QTcF or QTcB interval greater than or equal to 450 msec), respiratory (including active tuberculosis), history of jaundice, hepatic, renal, gastrointestinal, immunological, neurological (including auditory), endocrine, infectious, malignancy, psychiatric, history of convulsions or other abnormality (including head trauma).
7. Family history of sudden death or of congenital prolongation of the QT interval or any other clinical condition known to prolong the QT interval.
8. Known congenital prolongation of the QT-interval or any clinical condition known to prolong the QT interval.
9. History of symptomatic cardiac arrhythmias or with clinically relevant bradycardia.
10. Any predisposing cardiac conditions for arrhythmia such as severe hypertension, left ventricular hypertrophy (including hypertrophic cardiomyopathy) or congestive cardiac failure accompanied by reduced left ventricle ejection fraction.
11. Electrolyte disturbances, particularly hypokalaemia, hypocalcaemia or hypomagnesaemia.
12. Any treatment which can induce a lengthening of QT interval, such as:

    i. Antiarrhythmics (e.g. amiodarone, disopyramide, dofetilide, ibutilide, procainamide, quinidine, hydroquinidine, sotalol) ii. Neuroleptics (e.g. phenothiazines, sertindole, sultopride, chlorpromazine, haloperidol, mesoridazine, pimozide, or thioridazine) iii. Antidepressive agents, certain antimicrobial agents, including agents of the following classes macrolides (e.g. erythromycin, clarithromycin), fluoroquinolones (e.g. moxifloxacin, sparfloxacin), imidazole and triazole antifungal agents, and also pentamidine and saquinavir iv. Certain non-sedating antihistamines (e.g. terfenadine, astemizole, mizolastine), cisapride, droperidol, domperidone, bepridil, diphemanil, probucol, levomethadyl, methadone, vinca alkaloids, arsenic trioxide
13. Known history of hypersensitivity, allergic or adverse reactions to artemisinin containing compounds, piperaquine or naphthoquine or to any of the excipients contained in ARCO and Eurartesim.
14. Antimalarial treatment with different antimalarial drugs as follows i. Piperaquine-based compound, mefloquine, naphthoquine or sulphadoxine/pyrimethamine (SP) within the previous 3 months, ii. Amodiaquine or chloroquine within the previous 6 weeks, and with quinine, halofantrine, lumefantrine-based compounds and iii. Any other antimalarial treatment, antibiotics with antimalarial activity (including cotrimoxazole, tetracyclines, quinolones and fluoroquinolones, and azithromycin) or any herbal products, within the past 14 days
15. Have received an investigational drug within the past 6 weeks.
16. Liver function tests:

    i. If Total Bilirubin is normal, exclude the patient if liver function tests ASAT/ALAT ≥ 3xULN ii. If Total Bilirubin is > 1 and ≤ 1.5xULN, exclude the patient if ASAT/ALAT ≥2xULN.

    iii. Total Bilirubin >1.5xULN
17. Hb level below 9 g/dL.
18. Serum creatinine levels more than 2 times the upper limit of normal range in absence of dehydration. In case of important dehydration the creatinine should be lower than 2X ULN after oral/parenteral rehydration.
19. Female patients must be neither pregnant (as demonstrated by a negative serum pregnancy test) nor lactating, and must be willing to take measures not to become pregnant during the study period and safety follow-up period.
20. Previous participation in any malaria vaccine trial or received malaria vaccine in any other circumstance

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2014-01-07 (Actual); Primary Completion 2014-07-27 (Actual); Study Completion 2015-06-01 (Actual)

PRIMARY OUTCOMES:
Number of reported non serious and serious adverse events | Up to 6 Weeks

SECONDARY OUTCOMES:
12-lead ECG recordings: Heart rate, PR interval, QRS duration, QT interval, QTc (Fridericia and Bazett corrections), any T wave or U-wave morphology. | Holter recording will run continuously during 12 hours after the last dose of treatment
  For ARCO treatment arm (which will only receive a single dose of ARCO treatment), Holter recording will start 15 minutes before the dose of ARCO, and it will run continuously during 12 hours post dosing.
  For Eurartesim treatment arm (which will receive three daily doses of Euratertesim treatment), Holter recording will run for 15 minutes before the first dose, and then it will start again 15 minutes before the third dose (last dose) running continuously for 12 hours post dosing.

OTHER OUTCOMES:
Frequency of abnormal safety laboratory parameters (hematology, clinical chemistry, urinalysis and coagulation) and clinical parameters (blood pressure, pulse rate, temperature) | weekly up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Salim Abdulla, MD, PhD, Principal Investigator — Ifakara Health Institute
Locations (1):
- Ifakara Health Institute, Bagamoyo, Tanzania

REFERENCES:
- [Derived] Ali AM, Gausi K, Jongo SA, Kassim KR, Mkindi C, Simon B, Mtoro AT, Juma OA, Lweno ON, Gwandu CH, Bakari BM, Mbaga TA, Milando FA, Hamad A, Shekalaghe SA, Abdulla S, Denti P, Penny MA. Population Pharmacokinetics of Antimalarial Naphthoquine in Combination with Artemisinin in Tanzanian Children and Adults: Dose Optimization. Antimicrob Agents Chemother. 2022 May 17;66(5):e0169621. doi: 10.1128/aac.01696-21. Epub 2022 Apr 25. PMID 35465706